CLINICAL TRIAL: NCT05270447
Title: Short-Term Effects of Connective Tissue Massage After Hysterectomy: A Randomized Controlled Study
Brief Title: Short-Term Effects of Connective Tissue Massage After Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, hanife dogan, Assistant Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-KAEK-177
Record Dates: First submitted 2022-02-17; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Massage; Hysterectomy; Pain
MeSH Terms: conditions — Pain | interventions — Massage; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Total laparoscopic hysterectomy (TLH) Connetive tissue massage group (Experimental): Connective tissue massage+ routine care+ advising
  Interventions: Other: Massage and patient education; Behavioral: Routine care and advising
- Total laparoscopic hysterectomy (TLH) control group (Other): routine care+ advising
  Interventions: Behavioral: Routine care and advising
- Total abdominal hysterectomy (TAH) Connetive tissue massage group (Experimental): Connective tissue massage+ routine care+ advising
  Interventions: Other: Massage and patient education; Behavioral: Routine care and advising
- Total abdominal hysterectomy (TAH) control group (Other): routine care+ advising
  Interventions: Behavioral: Routine care and advising

INTERVENTIONS:
Other: Massage and patient education — Connective tissue manipulation: The patients were informed about CTM and its mechanism of action before starting the CTM application. CTM was performed by a trained physiotherapist as the patient was in a sitting position.
  Routine care and advising: In-bed activities were taught and recommended to the patients in both groups. In-bed activities; rotation, sitting on the bedside, breathing exercises, range of motion exercises for upper and lower extremities. In addition, hourly walking activities were recommended after the anesthetic effect wore off.
  Arms: Total abdominal hysterectomy (TAH) Connetive tissue massage group; Total laparoscopic hysterectomy (TLH) Connetive tissue massage group
Behavioral: Routine care and advising — Routine care and advising: In-bed activities were taught and recommended to the patients in both groups. In-bed activities; rotation, sitting on the bedside, breathing exercises, range of motion exercises for upper and lower extremities. In addition, hourly walking activities were recommended after the anesthetic effect wore off.

SUMMARY:
The aim of this study to investigate the effects of connective tissue massage (CTM) on pain, intestinal peristaltism and functionality after total laparoscopic (TLH) or abdominal hysterectomy (TAH). Patients who underwent TLH randomly group as TLH-CTM (n=15) and TLH control (n=16), and TAH randomly group as TAH-CTM (n=14) and TAH control (n=15). The postoperative daily monitoring sheet, Visual Analogue Scale (VAS), time of intestinal peristaltism employees to collect research data.

DETAILED DESCRIPTION:
Interventions In the control groups (TLH control and TAH control) only in-bed activities and walking recommendations will be given, and routine care (analgesics and wound care) applies. In addition, CTM applies in the CTM groups (TLH-CTM and TAH-CTM).

Connective tissue manipulation: The patients are informed about CTM and its mechanism of action before starting the CTM application. CTM is performed by a trained physiotherapist as the patient was in a sitting position. All posterior connective tissue areas (sacral, lumbar, lower thoracic, scapular, inter-scapular, and cervical) are stimulated. Both short and long strokes will use during the manipulation. Each stroke will repeate three times, first on the right and then on the left of all desired zones. All sessions will terminated with long bilateral strokes to the iliac crest and subcostal regions. During manipulation, the pad of the middle finger will be in contact with the patient's skin. Application will take approximately 30-35 minutes depending on the area treated. CTM will apply twice: at postoperative 3rd hour and after 24 hours.

Routine care and advising: In-bed activities will advice to the patients in both groups. In-bed activities are; rotation, sitting on the bedside, breathing exercises, range of motion exercises for upper and lower extremities. In addition, hourly walking activities are recommended after the anesthetic effect wore off. Vital signs (pulse rate, blood pressure, and respiratory rate) and body temperatures will evaluate regularly. The investigators, will determine the severity of severe pain with the VAS scale. According to the VAS scale, if the patient reports pain intensity between 7-10 out of 10, it means that she has severe pain. Patients will encourage for early ambulation. Initially, they walked 10-15 m inside their rooms and the amount of walking increased over time.

ELIGIBILITY:
Inclusion Criteria:

* volunteered to participate in the study,
* those who underwent benign abdominal or laparoscopic hysterectomy,
* who were stable at post-operative vital signs and those with no complications in the early postoperative period

Exclusion Criteria:

* they had oncological diseases,
* chronic pain history, prolapse,
* those who had previous abdominal surgery,
* those with known psychological problems. For the CTM groups,
* those with local infection (abscess etc.), open lesion/wound, scar tissue, edema, and hematoma in the lumbar region.

Ages: 41 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Pain score | Change from baseline to postoperative 2 days
  Visual analog scale was used to assess pain levels. The Visual analog scale, is a 10-cm horizontal line ranging from "No Pain-Score 0" to "Intolerable Pain-Score 10", where "0" indicates the absence of pain and "10" indicates the presence of very severe pain.Higher scores related with worse pain status.

SECONDARY OUTCOMES:
time of the first passage of flatus after the surgery | Two days
  time of the first passage of flatus after the surgery
the time of the first defecation after the surgery | Two days
  the time of the first defecation after the surgery
blood pressure before and after interventions | Two days
  Blood Pressure measurement before and after interventions (Systolic and Diastolic Pressure; in mmHg)
Heart Rate before and after interventions | Two days
  Heart Rate measurement before and after interventions (Beat per minute)
Respiratory rates before and after interventions | Two days
  Respiratory rates measurements (Breathing rate number per minute)
The difficulty levels of the patients during functional activities | Two days
  Assess with scoring to perceived difficulty. Patients scores difficulty in their activities of daily living 0 to 10. 0 means no difficulty, 10 means highest difficulty, very diffuculty performing activity

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No